CLINICAL TRIAL: NCT02488148
Title: Bikram Yoga and Vascular Health
Brief Title: The Effect of Bikram Yoga on Arterial Stiffness and Endothelial Function in Middle-Aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Stacy D. Hunter, University Affiliate, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-12-0043
Record Dates: First submitted 2015-06-24; First posted 2015-07-02 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hot yoga (Experimental): 3 hot yoga classes per week to be completed at local studios in Austin, TX.
  Interventions: Behavioral: Hot yoga
- Non-heated yoga (Experimental): 3 yoga classes to be completed at local studios in Austin, TX.
  Interventions: Behavioral: Non-heated yoga
- Control (No Intervention): Maintain usual activities for the 12-week duration of the study.

INTERVENTIONS:
Behavioral: Hot yoga — Subjects in the two intervention groups will complete the standard 26-posture Bikram yoga series in a studio heated at 41ºC (traditional environment) or in a studio at a room temperature of 22ºC whereas control group subjects will be instructed to maintain physical activity patterns for the 12-week study duration. Yoga classes will be held at the Pure Bikram Yoga downtown Austin location. Classes will be completed 3 times weekly for 12 weeks and consist of 90 minutes of yoga postures and breathing exercises.
  Other Names: Bikram yoga
  Arms: Hot yoga
Behavioral: Non-heated yoga — Subjects in the two intervention groups will complete the standard 26-posture Bikram yoga series in a studio heated at 41ºC (traditional environment) or in a studio at a room temperature of 22ºC whereas control group subjects will be instructed to maintain physical activity patterns for the 12-week study duration. Yoga classes will be held at the Pure Bikram Yoga downtown Austin location. Classes will be completed 3 times weekly for 12 weeks and consist of 90 minutes of yoga postures and breathing exercises.
  Arms: Non-heated yoga

SUMMARY:
Arterial stiffening and endothelial dysfunction are correlates of advancing age contributing to the decline in cardioprotection with age. Arterial stiffness and endothelial dysfunction are emerging risk factors for cardiovascular disease and predict future cardiac events. Vascular function has long been a target for lifestyle interventions with several studies showing improvements traditional exercise modes. However, the impact of yoga on vascular function remains elusive. This study will determine the effect of a 12-week Bikram yoga intervention on arterial stiffness and endothelial function in healthy, middle-aged adults.

The overall aim of this study is to determine the efficacy of Bikram yoga in improving vascular endothelial function and arterial distensibility in middle-aged adults with risk factors for coronary artery disease and to determine whether the heated environment plays a role in mediating these alterations in vascular function. The investigators propose to conduct a 12-week Bikram yoga intervention study in sedentary individuals in order to test the following hypotheses:

1. Bikram yoga will elicit reductions in arterial stiffness and enhancements in endothelial function in sedentary, middle-aged adults.
2. The postulated effects of Bikram yoga will be greater when practiced in a heated environment.

DETAILED DESCRIPTION:
Bikram yoga is a trademarked form of yoga in which a series of 26 yoga postures are performed in a heated (41ºC), humidified environment over a 90-minute period. Bikram yoga has rapidly gained popularity with approximately 300 studios currently operating in the U.S. The 90-minute session consists of pranayama (breathing), and standing, balancing, strengthening, and stretching asanas (postures) all performed in a sauna-like environment. Although this highly controlled style of yoga provides an optimal choice for interventional research studies, few studies have attempted to elucidate the health benefits associated with Bikram yoga.

Subjects will be randomly assigned to one of three groups: heated Bikram yoga (41ºC), room temperature Bikram yoga (22ºC), or control in which the participants will be instructed not to alter physical activity patterns. Collected data from this interventional study will be analyzed by ANOVA and/or ANCOVA with repeated measures. Pearson correlation coefficients will be used to examine associations between variables of interest. A significance level of p<0.05 will be employed to determine statistical significance.

A total of 80 sedentary (<2 days of physical activity weekly) male and female adults between the ages of 40 and 60 years will be recruited and studied. Twenty subjects in each group will complete 12 weeks of Bikram yoga at room temperature (22ºC), Bikram yoga in a heated environment (41ºC), or a control period during which participants will be instructed not to alter physical activity levels. Based on a previous study competed by the investigators which employed Bikram yoga as an intervention, a dropout rate of 25% is anticipated. Therefore, as the goal of the investigators is to have a minimum of 60 subjects (20 per group) complete the 12-week intervention, the investigators will recruit and enroll 80 subjects.

Once participants report to the laboratory, height and weight will be measured and a finger prick will be performed. Body composition will then be measured via dual energy x-ray absorptiometry scan.

Endothelial function will be measured non-invasively via flow-mediated dilation. This technique involves ultrasound imaging of the upper arm to obtain an image of the brachial artery. Once baseline images are acquired, a cuff placed around the forearm will be inflated for 5 minutes. More images will be acquired after the cuff is deflated and the images will be analyzed to determine the percent change in arterial diameter from baseline.

Arterial stiffness will be measured using pulse wave velocity. Tonometric sensors will be placed on the carotid and femoral pulse sites and blood pressure cuffs placed on the arms and ankles to determine brachial and tibial arterial blood pressure. The distance between the carotid and femoral pulse sites will be measured and pulse wave velocity will be determined as distance traveled divided by the time between the initiation of the carotid and femoral pulses.

ELIGIBILITY:
Inclusion Criteria:

* A total of 80 sedentary (<2 days of physical activity weekly) male and female adults between the ages of 40 and 60 years will be recruited and studied.

Exclusion Criteria:

* pregnancy (if the subject is unsure about her status, a simple testing kit will be made available to the subject)
* Uncontrolled hypertension (blood pressure >160/100 mmHg while on hypertensive medications)
* Infection within the previous 4 weeks
* Having adrenal or endocrine tumors
* Renal disease
* Prior myocardial infarction (heart attack)
* Known coronary artery disease
* Personal history of stroke
* Heart failure
* Cardiac arrhythmias
* Chronic obstructive pulmonary disease
* Personal history of psychosis
* Diabetes
* Having a body mass index ≥35 kg/m2
* Recent chest pain or dyspnea
* Orthopedic limitations that prevent them from being able to perform the yoga postures
* Heat intolerance
* Having undergone a barium test within the previous two weeks
* Having had a nuclear medicine scan or injection with x-ray dye within the previous week.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 12 weeks
  Endothelial function will be measured non-invasively via flow-mediated dilation at baseline and after 12 weeks. This technique involves ultrasound imaging of the upper arm to obtain an image of the brachial artery. Once baseline images are acquired, a cuff placed around the forearm will be inflated for 5 minutes. More images will be acquired after the cuff is deflated and the images will be analyzed to determine the percent change in arterial diameter from baseline.
Arterial stiffness (pulse wave velocity) | 12 weeks
  Arterial stiffness will be measured using pulse wave velocity at baseline and 12 weeks. Tonometric sensors will be placed on the carotid and femoral pulse sites and blood pressure cuffs places on the arms and ankles to determine brachial and tibial arterial blood pressure. The distance between the carotid and femoral pulse sites will be measured and pulse wave velocity will be determined as distance traveled divided by the time between the initiation of the carotid and femoral pulses.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Hunter, PhD, Principal Investigator — University of Texas
Locations (1):
- Cardiovascular Aging Research Laboratory, Austin, Texas, United States